CLINICAL TRIAL: NCT05183750
Title: Ankle Pain and Orientation After High Tibial Osteotomy as a Treatment of Medial Compartment Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Lotfy Saber Mohammed, Specialist of Orthopedic and Trauma Surgery, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-21-12-18
Record Dates: First submitted 2021-12-17; First posted 2022-01-11 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Investigate the Change in the Weight-bearing-line (WBL) Ratio of the Ankle Joint and Ankle Joint Line Orientation After HTO

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult with isolated medial compartmental knee osteoarthtitis (Other)
  Interventions: Procedure: High tibial osteotomy

INTERVENTIONS:
Procedure: High tibial osteotomy — Opening wedge high tibial osteotomy will be done according to the measurement preoperatively and fixation will be by plate and screws.

SUMMARY:
Changes in demographics and physical activities of the young population have increased the number of patients with medial unicompartmental knee osteoarthritis (OA) requiring surgical intervention.

High tibial osteotomy (HTO) have shown good clinical results in restoring lower extremity alignment, reducing pain, and improving knee function in patients with moderate-to-severe knee osteoarthritis and genu varum deformity.

The aim of this study is to evaluate the relation between correction of the malalignment of the knee and ankle pain and orientation in patient of medial compartment knee osteoarthritis using high tibial osteotomy by recent reports concerning the indications, functional outcomes and complication.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is highly prevalent worldwide. It is a leading cause of musculoskeletal disability and associated with activity limitation, working disability and reduced quality of life.

Osteoarthritis can affect any synovial joint in the body, however it occurs most often in weight-bearing joints, with the knee being one of the most commonly affected. Progressive loss of hyaline articular cartilage is often considered the hallmark of the disease. Within the tibiofemoral joint; articular cartilage degradation is most prevalent in the medial compartment.

Changes in demographics and physical activities of the young population have increased the number of patients with medial unicompartmental knee osteoarthritis (OA) requiring surgical intervention.

High tibial osteotomy (HTO) have shown good clinical results in restoring lower extremity alignment, reducing pain, and improving knee function in patients with moderate-to-severe knee osteoarthritis and genu varum deformity.

Prior to the development of total knee arthroplasty (TKA) as a reliable procedure in the 1980s, high tibial osteotomy (HTO) was the most common surgical treatment for varus gonarthrosis.

HTO may influence the alignment and function of the ankle joint. In the case of greater varus deformity where the preoperative talar tilt was increased medial to the ankle or the postoperative correction angle was large, the incidence of arthritis in the ankle joint rose Therefore, it is possible for realignment procedures in the knee HTO to affect ankle joint alignment and ankle symptoms.

Assessment of change in the weight-bearing-line (WBL) ratio of the ankle joints would provide a theoretical basis for post-operative ankle joint pain and osteoarthritis progression after knee arthroplasty or HTO.

The aim of this study is to evaluate the relation between correction of the malalignment of the knee and ankle pain and orientation in patient of medial compartment knee osteoarthritis using high tibial osteotomy by recent reports concerning the indications, functional outcomes and complication .

So this study aimed to investigate the change in the weight-bearing-line (WBL) ratio of the ankle joint and ankle joint line orientation after HTO in patients with genu varum deformity.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic medial unicompartment knee arthritis
* Active patients younger than 55 years
* Good range of motion (ROM) .
* Intact lateral compartment

Exclusion Criteria:

* Combined medial and lateral arthrosis.
* Markedly decreased knee range of motion (arc of motion 10°).
* Ligamentous instability.
* Severe joint destruction (≥Ahlback grade III).
* ≥55 years of age.
* Advanced patellofemoral arthritis.
* Rheumatoid arthritis.
* Structural lower extremity deformities.
* Previous operation at knee joint.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Ankle pain (visual analogue score) | 1year post operative follow up
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores represents a continuum between no pain 0 and worst pain 10.
Coronal alignment of the ankle | 1year post operative follow up
  Tibial plafond inclination (TPI) (2) Talar inclination (TI) (3) Talar tilt (TT)and (4) Lateral distal tibial angle (LDTA)
coronal plane correction | 1year post operative follow up
  hip-knee-ankle (HKA) angle, medial proximal tibial angle (MPTA), and knee-tibial plafond angle (KTPA)

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag univeristy- Faculty of medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kijowski R, Blankenbaker D, Stanton P, Fine J, De Smet A. Arthroscopic validation of radiographic grading scales of osteoarthritis of the tibiofemoral joint. AJR Am J Roentgenol. 2006 Sep;187(3):794-9. doi: 10.2214/AJR.05.1123. PMID 16928947
- [Background] Lee JH, Jeong BO. Radiologic changes of ankle joint after total knee arthroplasty. Foot Ankle Int. 2012 Dec;33(12):1087-92. doi: 10.3113/FAI.2012.1087. PMID 23199858
- [Background] Ducat A, Sariali E, Lebel B, Mertl P, Hernigou P, Flecher X, Zayni R, Bonnin M, Jalil R, Amzallag J, Rosset P, Servien E, Gaudot F, Judet T, Catonne Y. Posterior tibial slope changes after opening- and closing-wedge high tibial osteotomy: a comparative prospective multicenter study. Orthop Traumatol Surg Res. 2012 Feb;98(1):68-74. doi: 10.1016/j.otsr.2011.08.013. Epub 2012 Jan 12. PMID 22244250
- [Background] Gaasbeek R, Welsing R, Barink M, Verdonschot N, van Kampen A. The influence of open and closed high tibial osteotomy on dynamic patellar tracking: a biomechanical study. Knee Surg Sports Traumatol Arthrosc. 2007 Aug;15(8):978-84. doi: 10.1007/s00167-007-0305-0. Epub 2007 May 5. PMID 17483931
- [Background] JACKSON JP, WAUGH W. Tibial osteotomy for osteoarthritis of the knee. J Bone Joint Surg Br. 1961 Nov;43-B:746-51. doi: 10.1302/0301-620X.43B4.746. No abstract available. PMID 14036496
- [Background] Lustig S, Scholes CJ, Costa AJ, Coolican MJ, Parker DA. Different changes in slope between the medial and lateral tibial plateau after open-wedge high tibial osteotomy. Knee Surg Sports Traumatol Arthrosc. 2013 Jan;21(1):32-8. doi: 10.1007/s00167-012-2229-6. Epub 2012 Oct 4. PMID 23052121